CLINICAL TRIAL: NCT01065701
Title: Comparison of Two Doses of Intranasal Dexmedetomidine as Premedication in Children - a Double-blinded Randomized Controlled Trial
Brief Title: Comparison of Two Doses of Intranasal Dexmedetomidine as Premedication in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, YUEN, Vivian Man-ying, Dr., The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: InDex3
Record Dates: First submitted 2010-02-07; First posted 2010-02-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Patient Between 1-8 Years Old Undergoing Elective Surgery at Queen Mary Hospital
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1mcg/kg (Active Comparator): 1mcg/kg intranasal dexmedetomidine administered 45 minutes befoe anesthesia induction
  Interventions: Drug: Dexmedetomidine
- 2mcg/kg (Active Comparator): 2mcg/kg intranasal dexmedetomidine given 45 minutes prior to anesthetic induction
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Intranasal dexmedetomidine is given as premedication prior to induction of anesthesia

SUMMARY:
Intranasal dexmedetomidine has shown to be an effective sedative when used prior to anaesthetic induction as premedication. 1mcg/kg intranasal dexmedetomidine was used in previous study and it produced satisfactory sedation in more than 50% of the children at the time of anaesthetic induction with no adverse effect. In this study we aim to compare 1mcg/kg with 2mcg/kg intranasal dexmedetomidine in children. We expect more children would attain satisfactory sedation prior to anaesthetic induction when higher dose is used.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-12 years old
* American Society of Anesthesiologists (ASA) 1-2
* Elective surgery
* Children with autism or pervasive personality disorder

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) 3-5
* Allergy or hypersensitive reaction to dexmedetomidine
* Known cardiac arrhythmia or congenital heart disease
* Mentally disabled

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
proportion of children attained satisfactory sedation | one hour

SECONDARY OUTCOMES:
time to onset of sedation | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Vivian M Yuen, MBBS, Principal Investigator — Associate Consultant, Queen Mary Hospital
Locations (1):
- QUeen Mary Hospital, Hong Kong, Hong Kong